CLINICAL TRIAL: NCT03675919
Title: The Telemedical Lifestyle Intervention Program TeLIPro (TeLIPro Health Program - Active With Diabetes)
Brief Title: TeLIPro Health Program - Active With Diabetes
Acronym: TeLIPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: AOK Rheinland/Hamburg (Industry); German Institute for Telemedicine and Health Promotion (Other); German Diabetes Center (Other)
Responsible Party: Principal Investigator, Stephan Martin, Director, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TeLIPro
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will be provided a scale, a step counter as well as access to the online portal and will remain in routine care.
  Interventions: Device: Scale; Device: Step counter; Other: Access to the online portal
- TeLIPro group (Experimental): The TeLIPro group will be provided a scale, a step counter, a blood glucose meter with test stripes as well as access to the online portal and will get telemedical coaching.
  Interventions: Device: Scale; Device: Step counter; Device: Blood glucose meter with test stripes; Other: Access to the online portal; Other: Telemedical coaching

INTERVENTIONS:
Device: Scale — self-monitoring of body weight; with automatic data transfer into the personalized and secured online portal
Device: Step counter — self-monitoring of physical activity; with automatic data transfer into the personalized and secured online portal
Device: Blood glucose meter with test stripes — self-monitoring of blood glucose; with automatic data transfer into the personalized and secured online portal
  Arms: TeLIPro group
Other: Access to the online portal — self-monitoring of health parameters
Other: Telemedical coaching — regular telephone calls providing information about T2DM, healthy lifestyle, low-carbohydrate diet and physical activity
  Arms: TeLIPro group

SUMMARY:
In a randomized-controlled trial the hypothesis should be tested that the Telemedical Lifestyle Intervention Program TeLIPro could significantly improve HbA1c (primary outcome), body weight and composition, cardiovascular risk factors, quality of life, eating behavior, and medication demand (secondary outcomes) in type 2 diabetes mellitus (T2DM) patients.

DETAILED DESCRIPTION:
T2DM patients, assured at the health insurance AOK Rhineland / Hamburg will be randomized into two parallel groups. In addition to routine care both groups will be provided a scale as well as a step counter and access to a secured online portal. The TeLIPro group will additionally got a glucose meter with test stripes fpr self-monitoring of blood glucose and telemedical coaching.

Participants of both groups will enter their anthropometric and metabolic data into a database on quarterly basis. In addition, the costs for diabetes-specific treatment, inpatient and outpatient treatment costs and drug costs will be analyzed on the basis of the routine data of the AOK Rhineland / Hamburg.

Patient preference for type 2 diabetes intervention will be recorded using Discrete Choice Experiment (DCE) questionnaires at the beginning of the program and at the end of the intervention. As part of the development and validation of the DCE, focus groups are used to determine the DCE attributes. In addition, focus groups should also be used during the data collection in order to obtain additional information on patient preferences by means of qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* body mass index of et least 27 kg/m2

Exclusion Criteria:

* acute infections
* chronic diseases other than type 2 diabetes and hypertension (e.g., cancer, chronic obstructive pulmonary disease, asthma, dementia, chronic gut diseases, psychoses, liver cirrhosis, macronephropathy/nephropathy, kidney insufficiency with glomerular filtration rate <30 ml/min/1.73 m2)
* acute chemotherapy or chronic cortisol treatment
* smoking cessation for <3 months and/or planned smoking cessation during study
* pregnancy or breast-feeding

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1163 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
HbA1c change | 12 months
  estimated treatment difference between groups of HbA1c change (in T2DM patients with diabetes duration of ≥ 5 years)
remission rate | 12 months
  number of participants with an HBA1c <6.5% (in T2DM patients with diabetes duration of < 5 years)

SECONDARY OUTCOMES:
fasting blood glucose change | 12 months
  estimated treatment difference between groups of fasting blood glucose change
weight change | 12 months
  estimated treatment difference between groups of weight change
body mass index change | 12 months
  estimated treatment difference between groups of body mass index change
systolic blood pressure change | 12 months
  estimated treatment difference between groups of systolic blood pressure change
diastolic blood pressure change | 12 months
  estimated treatment difference between groups of diastolic blood pressure change
total cholesterol change | 12 months
  estimated treatment difference between groups of total cholesterol change
high-density lipoprotein (HDL) cholesterol change | 12 months
  estimated treatment difference between groups of high-density lipoprotein (HDL) cholesterol change
low-density lipoprotein (LDL) cholesterol change | 12 months
  estimated treatment difference between groups of low-density lipoprotein (LDL) cholesterol change
triglyceride change | 12 months
  estimated treatment difference between groups of triglyceride change
number of steps | 12 months
  estimated treatment difference between groups of number of steps
antidiabetic medication change | 12 months
  estimated treatment difference between groups of antidiabetic medication change
diabetes-specific treatment costs | 12 months
  estimated treatment difference between groups of diabetes-specific treatment costs
inpatient costs | 12 months
  estimated treatment difference between groups of inpatient costs
outpatient costs | 12 months
  estimated treatment difference between groups of outpatient costs

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Altpeter, Study Chair — Deutsches Institut für Telemedizin und Gesundheitsförderung; Sibel Altin, Study Chair — AOK Rheinland/Hamburg; Andrea Icks, PhD, Study Chair — Deusches Diabetes Zentrum
Locations (1):
- West German Centre of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No